CLINICAL TRIAL: NCT01675011
Title: Safety and Efficacy of Embozene Microspheres for Uterine Fibroid Embolization Compared to Embosphere for Symptomatic Relief From Uterine Fibroids
Brief Title: Embozene Microspheres for Uterine Fibroid Embolization (UFE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-001
Record Dates: First submitted 2012-08-25; First posted 2012-08-29 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Embozene® Microspheres (Experimental): Uterine Fibroid Embolization (UFE)will be used to treat the fibroids. The procedure involves injecting embolizing particles into the uterine artery which causes the fibroid to shrink.
  Interventions: Device: Embozene® Microspheres
- Embosphere® (Active Comparator): Uterine Fibroid Embolization (UFE)will be used to treat the fibroids. The procedure involves injecting embolizing particles into the uterine artery which causes the fibroid to shrink.
  Interventions: Device: Embosphere®

INTERVENTIONS:
Device: Embozene® Microspheres
  Arms: Embozene® Microspheres
Device: Embosphere®
  Arms: Embosphere®

SUMMARY:
This is a randomized, prospective, multi-center study of 225 female subjects age 30-50 years with symptoms from uterine fibroids. All subjects will be followed for a total of thirty-six (36) months following uterine fibroid embolization.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent and must sign the Institutional Review Board approved Informed Consent Form.
* Pre-menopausal women age 30-50 years at time of enrollment
* Have been selected forUterine Fibroid Embolization (UFE) prior to entry to the study.

Exclusion Criteria:

* Patient has a history of pelvic malignancy
* Patient has an abnormal Pap smear within 12 months of the planned Uterine Fibroid Embolization procedure
* Patient with coexisting condition that might explain abnormal bleeding (including endometrial hyperplasia and adenomyosis) or pelvic pain (including endometriosis and ovarian cysts).
* Is at substantial risk for the need of organ transplantation, such as renal insufficiency.
* Patient has evidence of current or recent pelvic inflammatory disease or uterine infection.
* Patient with a severe contrast allergy or renal insufficiency that would represent a contradiction to the administration of iodine-based contrast agents.
* Patients unable to comply with the follow-up requirements of the study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Albany Medical Center, Albany, New York
  - North Shore LIJ Medical Center, New Hyde Park, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 patients screened and 4 randomized.
Groups:
- Embozene® Microspheres: Uterine Fibroid Embolization (UFE)will be used to treat the fibroids. The procedure involves injecting embolizing particles into the uterine artery which causes the fibroid to shrink.
  Embozene® Microspheres
- Embosphere®: Uterine Fibroid Embolization (UFE)will be used to treat the fibroids. The procedure involves injecting embolizing particles into the uterine artery which causes the fibroid to shrink.
  Embosphere®
Period: Overall Study
Arm/Group | Embozene® Microspheres | Embosphere®
Started | 3 | 1
Completed | 0 | 0
Not Completed | 3 | 1
Not completed — Trial terminated by Sponsor | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Embozene® Microspheres | Embosphere® | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 45 [40 to 49] | 45 [45 to 45] | 45 [40 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint
Description: The primary effectiveness endpoint for this clinical trial is the proportion of subjects who have success, defined as 50% menstrual blood loss (MBL) reduction or less than 80 ml of MBL per cycle, evaluated by the Alkaline Hematin (AH) method, at 12 months.
Time Frame: 12 Months post study procedure
Population: The study was terminated due to inadequate enrollment; no patients completed the 12 month visit.
Arm/Group | Embozene® Microspheres | Embosphere®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 through 6 months.
Arm/Group | Embozene® Microspheres | Embosphere®
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Embozene® Microspheres (N=3) | Embosphere® (N=1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to insufficient enrollment, therefore formal statistical analyses were not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No